CLINICAL TRIAL: NCT00605722
Title: A Single Arm, Open Label Study of First Line Treatment With Tarceva Plus Avastin on Progression-free Survival in Patients With Advanced or Metastatic Liver Cancer
Brief Title: A Study of Tarceva (Erlotinib) and Avastin (Bevacizumab) in Patients With Advanced or Metastatic Liver Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21213
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-06

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Bevacizumab; Erlotinib Hydrochloride

ARMS (1):
- bevacizumab + erlotinib (Experimental): Participants received bevacizumab (Avastin) 5 mg/kg intravenous (iv) on day 1 of each 2 week cycle plus erlotinib (Tarceva) 150 mg orally once a day until disease progression or unmanageable toxicity.
  Interventions: Drug: bevacizumab (Avastin); Drug: erlotinib (Tarceva)

INTERVENTIONS:
Drug: bevacizumab (Avastin) — 5 mg/kg iv on day 1 of each 2 week cycle.
Drug: erlotinib (Tarceva) — 150 mg orally (po) daily.

SUMMARY:
This single arm study evaluated the efficacy and safety of a combination of Tarceva and Avastin in patients with advanced or metastatic liver cancer. Patients were treated with Tarceva 150 mg po daily plus Avastin 5 mg/kg intravenous (iv) every 2 weeks. The anticipated time on study treatment was until disease progression, and the target sample size was <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, ≥ 18 years of age;
* advanced or metastatic liver cancer;
* ≥ 1 measurable lesion, not previously treated with local therapy within 4 weeks of enrollment.

Exclusion Criteria:

* prior or concomitant systemic anti-cancer treatment for advanced disease;
* patients at high risk of variceal bleeding;
* clinically significant cardiovascular disease;
* major surgery, open biopsy, or significant traumatic injury within 4 weeks of study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Manila, Philippines
- Seoul, South Korea
- Taiwan (3):
  - Kueishan
  - Tainan
  - Taipei

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab + Erlotinib
Started | 51
Completed | 0 (Completed=Completed Treatment.)
Not Completed | 51
Not completed — Adverse Event | 6
Not completed — Insufficient therapeutic response | 44
Not completed — Failure to return | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab + Erlotinib
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (14.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 44

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-free Survival (PFS)
Description: Percentage of participants who were alive and without documented progressive disease 16 weeks after their first dose of study drug. Diagnosis of Progressive Disease was made by objective criteria (RECIST criteria) on the target lesion(s), or by documenting, with Computerised Tomography/Magnetic Resonance Imaging (CT/MRI) scans, the presence of newly occurring lesion(s) arising outside the scanned areas of the target lesions. PD required at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Week 16
Population: Intent-to-treat population included all participants who received study drug. Participants who had neither progressed nor died at the time of study completion or who were lost to follow-up were censored at the date of the last tumor assessment or last follow up for progression of disease.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Erlotinib
Number analyzed (Participants) | 51
percentage of participants | 35.3 [22.4 to 49.9]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with Complete Response (CR) or Partial Response (PR). Analysis of tumor response was based on the best overall response according to Response Evaluation Criteria in Solid Tumors (RECIST), which was defined as the best response recorded from the start of trial treatment until disease progression/recurrence (or death), taking as reference for progressive disease (PD) the smallest measurements recorded since the treatment started. CR was defined as the disappearance of all target lesions; for non-target lesions disappearance of lesions and normal tumour marker levels. PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, using as reference the Baseline sum LD. PD required at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Event driven (median follow-up 12 months)
Population: Intent-to-treat population included all participants who received study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Erlotinib
Number analyzed (Participants) | 51
percentage of participants
  Complete Response | 0.0 [0.0 to 7.0]
  Partial Response | 5.9 [1.2 to 16.2]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease Control Rate was defined as the percentage of participants with Complete Response (CR), Partial Response (PR) or Stable Disease (SD) for at least 8 weeks by Response Evaluation Criteria in Solid Tumours (RECIST). CR was defined as the disappearance of all target lesions; for non-target lesions disappearance of lesions and normal tumour marker levels. PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, using as reference the Baseline sum LD. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started; for non-target lesions persistence of one or more non-target lesion(s) and/or maintenance of tumour marker level above the normal limits.
Time Frame: Event driven (median follow-up 12 months)
Population: Intent-to-treat population included all participants who received study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bevacizumab + Erlotinib
Number analyzed (Participants) | 51
Percentage of participants | 52.9 [38.5 to 67.1]

4. Secondary Outcome: Time to Tumor Progression
Description: Time to tumor progression was defined as the time period in months from the start of study drug treatment to disease progression. Progressive disease required at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Event driven (median follow-up 12 months)
Population: Intent-to-treat population included all participants who received study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Erlotinib
Number analyzed (Participants) | 51
Months | 2.9 [1.8 to 5.3]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time period in months from the start of study drug treatment to the first of either progression or death. Progressive disease required at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Event driven (median follow-up 12 months)
Population: Intent-to-treat population included all participants who received study drug. Participants were censored at the last follow-up visit.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Erlotinib
Number analyzed (Participants) | 51
months | 2.9 [1.8 to 4.8]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time period in months from the start of study drug treatment to death.
Time Frame: Event driven (median follow-up 12 months)
Population: Intent-to-treat population included all participants who received study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Erlotinib
Number analyzed (Participants) | 51
months | 10.7 [7.4 to NA] — Kaplan-Meier estimate; Confidence Interval (CI) was not estimated due to the small number of participants with events.

7. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study and laboratory or clinical tests that resulted in a change in treatment or discontinuation from study drug were reported as adverse events. A SAE was any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: Up to 107 Weeks
Population: Safety population included all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Erlotinib
Number analyzed (Participants) | 51
participants
  Serious Adverse Events | 19
  Adverse Events | 51

ADVERSE EVENTS:
Time Frame: Up to 107 weeks
Arm/Group | Bevacizumab + Erlotinib
Serious Adverse Events (participants affected / at risk) | 19/51
Other Adverse Events (participants affected / at risk) | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Erlotinib (N=51)
Anemia (Blood and lymphatic system disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2
Tumor associated fever (General disorders) | 2
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastric varices hemorrhage (Gastrointestinal disorders) | 1
Melena (Gastrointestinal disorders) | 1
Peptic ulcer (Gastrointestinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Anal abscess (Infections and infestations) | 1
Bacteremia (Blood and lymphatic system disorders) | 1
Enterobacter infection (Infections and infestations) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Hepatic failure (Renal and urinary disorders) | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Tumor pain (General disorders) | 1
Inappropriate anti-diuretic hormone secretion (Endocrine disorders) | 1
Pyrexia (General disorders) | 1
Transaminase increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hepatic encephalopathy (Hepatobiliary disorders) | 1
Bleeding varicose vein (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Erlotinib (N=51)
Rash (Skin and subcutaneous tissue disorders) | 36
Acne (Skin and subcutaneous tissue disorders) | 22
Palmer-Plantar erythrodysaesthesis syndrome (Skin and subcutaneous tissue disorders) | 11
Pruritus (Skin and subcutaneous tissue disorders) | 11
Alopecia (Skin and subcutaneous tissue disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 6
Diarrhea (Gastrointestinal disorders) | 26
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 8
Stomatitis (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 6
Gastric ulcer (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 4
Gingival bleeding (Gastrointestinal disorders) | 3
Melena (Gastrointestinal disorders) | 3
Mouth ulceration (Gastrointestinal disorders) | 3
Varices esophageal (Gastrointestinal disorders) | 3
Pyrexia (General disorders) | 13
Fatigue (General disorders) | 9
Edema peripheral (General disorders) | 5
Asthenia (General disorders) | 4
Chest pain (General disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 5
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Paronychia (Infections and infestations) | 10
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 20
Weight decreased (Investigations) | 9
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 4
Dizziness (Nervous system disorders) | 7
Dysgeusia (Nervous system disorders) | 3
Proteinuria (Renal and urinary disorders) | 6
Hematuria (Renal and urinary disorders) | 3
Insomnia (Psychiatric disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 3
Anemia (Blood and lymphatic system disorders) | 6
Hypertension (Vascular disorders) | 6
Hyperbilirubinemia (Hepatobiliary disorders) | 5
Cataract (Eye disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.